CLINICAL TRIAL: NCT00930085
Title: Evaluation of Predictive Proteic Profile on Mortality in the Acute Phase of Septic Shock in Cancer Patients
Acronym: PROTEOHSEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PROTEOHSEPS/IPC 2005-011
Record Dates: First submitted 2009-06-22; First posted 2009-06-30 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Sepsis; Septic Shock; Cancer
Keywords: sepsis; septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic; Neoplasms | interventions — Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SELDI-TOF MS (Experimental): The proteic profiling is performed by SELDI-TOF mass spectroscopy.
  Interventions: Other: SELDI-TOF MS for plasmatic proteic profile

INTERVENTIONS:
Other: SELDI-TOF MS for plasmatic proteic profile — An extra blood sample is required to determine the plasmatic proteic profile used to identify one or several signatures which are correlated to the clinical evolution (mortality at D30).

SUMMARY:
The mortality induced by infections in onco-hematological patients is abnormally high at the acute phase of septic shock. Consequently, it is important to detect the population with a high risk of short term mortality among patients with a septic shock. The aim of this study is the evaluation of predictive proteic profile on the short term mortality in the acute phase of septic shock in cancer patients.

DETAILED DESCRIPTION:
Method: Monocentric prospective study with diagnostic and prognostic expectations.

Primary objective:

Identification and characterization of early proteic biomarkers predictive of short term mortality in cancer patients with septic shock.

Secondary objective:

Research of clinical and biological prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient from oncology or hematology with a septic shock
* Patient aged 18 years and older
* Inclusion within the 24 hours of the septic shock in the intensive care unit
* Signed consent according to the emergency reglementation

Exclusion Criteria:

* Pregnancy, breast feeding
* Patient with decision of care limitation
* Patient with legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Identification and characterization of early proteic biomarkers predictive of short term mortality in cancer patients with septic shock. | 1 month

SECONDARY OUTCOMES:
Research of clinical and biological prognostic factors. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Djamel MOKART, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr